CLINICAL TRIAL: NCT06487559
Title: A Phase 1b Study to Evaluate the Safety and Pharmacokinetics of Livmoniplimab in Combination With Budigalimab in Chinese Subjects With Locally Advanced or Metastatic Child-Pugh A Hepatocellular Carcinoma Who Have Progressed After a First-Line Regimen That Includes an Immune Checkpoint Inhibitor
Brief Title: A Study to Assess the Adverse Events and How Intravenously Infused Livmoniplimab in Combination With Budigalimab Moves Through the Bodies of Adult Chinese Participants With Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-695
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma (HCC); Livmoniplimab; ABBV-151; budigalimab; ABBV-181
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1: Cohort 1 Livmoniplimab + Budigalimab Dose A (Experimental): Participants will receive livmoniplimab Dose A in combination with budigalimab every 3 weeks for approximately 2 years.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Stage 2: Cohort 2 Livmoniplimab + Budigalimab Dose B (Experimental): Participants will receive livmoniplimab Dose B in combination with budigalimab every 3 weeks for approximately 2 years.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab

INTERVENTIONS:
Drug: Livmoniplimab — Intravenous infusion
  Other Names: ABBV-151
Drug: Budigalimab — Intravenous infusion
  Other Names: ABBV-181

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cancer worldwide and a leading cause of cancer-related death. The majority of participants first presenting with HCC have advanced unresectable or metastatic disease. The purpose of this study is to assess adverse events and how livmoniplimab in combination with budigalimab moves through the body in adult Chinese participants with Locally Advanced or metastatic Child-Pugh A Hepatocellular Carcinoma (HCC).

Livmoniplimab is an investigational drug being developed for the treatment of HCC. There are 2 stages to this study. Stage 1 is a safety run-in. There are 2 treatment arms in stage 1 and participants will receive escalating doses of Livmoniplimab in combination with budigalimab (fixed dose). Stage 2 is dose expansion. There are 2 treatment arms in stage 2 and participants will receive Livmoniplimab in combination with budigalimab in multiple doses. Approximately 20 adult participants will be enrolled in the study across 15 sites in China.

In part 1 (dose escalation), participants will be intravenously infused with escalating doses of livmoniplimab in combination with budigalimab every 3 weeks. In part 2 (dose expansion), participants will be intravenously infused with livmoniplimab in combination with budigalimab in multiple doses every 3 weeks. The estimated duration of the study is up to 2 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC
* Child-Pugh A
* Barcelona Clinic Liver Cancer stage B or C
* Eastern Cooperative Oncology Group (ECOG) Perfromance Status of 0-1
* Received an immune checkpoint inhibitor in 1L HCC treatment regimen
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases as outlined in the protocol.
* History of malignancy other than HCC within 5 years prior to screening, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%).
* History of autoimmune, immune deficiency, or inflammatory disorders including, but not limited to, inflammatory bowel disease, systemic lupus erythematosus, sarcoidosis, Wegener syndrome, rheumatoid arthritis, antiphospholipid antibody syndrome, Guillain-Barre syndrome, or multiple sclerosis
* History of clinically significant conditions such as but not limited to the following: renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, pulmonary, or hepatic disease within the last 6 months that in Investigator's opinion, would adversely affect the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AE) | Up to Approximately 2 Years
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Number of Participants with Dose-Limiting Toxicities (DLT) | Up to Approximately 2 Years
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Maximum Plasma Concentration (Cmax) of Livmoniplimab and Budigalimab | Up to Approximately 2 Years
  Maximum Plasma Concentration (Cmax) of livmoniplimab and Budigalimab
Area Under the Serum Concentration Versus Time Curve (AUC) of Livmoniplimab and Budigalimab | Up to Approximately 2 Years
  AUC of livmoniplimab and Budigalimab

SECONDARY OUTCOMES:
Best Overall Response (BOR) for Participants with Confirmed CR/PR per RECIST v1.1 | Up to Approximately 2 Years
  Defined as achieving either confirmed CR or confirmed PR per RECIST v1.1 as assessed by the investigator.
Duration of response (DOR) for Participants with Confirmed CR/PR | Up to Approximately 2 Years
  Defined as the time from the participant's initial response (CR or PR) to the first occurrence of radiographic progression per RECIST v1.1 as determined by the investigator or death from any cause.
Progression-free survival (PFS) | Up to Approximately 2 Years
  Defined as the time from the participant's first dose of study drug until radiographic progression per RECIST v1.1 as determined by the investigator or death from any cause, whichever occurs first.
Overall survival (OS) | Up to Approximately 2 Years
  Defined as the time from the participant's first dose of study drug until death from any cause.
Antidrug Antibody (ADA) | Up to Approximately 2 Years
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antidrug Antibody (nADA) | Up to Approximately 2 Years
  Incidence and concentration of neutralizing anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- China (11):
  - Beijing Youan Hospital, Capital Medical University -No differernce with previous /ID# 261928, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University /ID# 262443, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 262092, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 262091, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital /Id# 262070, Harbin, Heilongjiang
  - Henan Cancer Hospital /ID# 262098, Zhengzhou, Henan
  - Hubei Cancer Hospital /ID# 262030, Wuhan, Hubei
  - The Second Affiliated Hospital of Nanchang University /ID# 262085, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute /ID# 268023, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University /ID# 262135, Shanghai, Shanghai Municipality
  - Zhejiang Cancer hospital /ID# 262046, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-695